CLINICAL TRIAL: NCT00479219
Title: A Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSI-953 in Blood and Cerebrospinal Fluid, When Administered Orally to Healthy Young Subjects and Patients With Alzheimer Disease
Brief Title: Study Evaluating GSI-953 in Healthy Young and Alzheimer's Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3183A1-103
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: GSI-953
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSI-953
  Arms: A
Other: Placebo
  Arms: B

SUMMARY:
To assess the pharmacodynamics (PD) of biomarkers amyloid beta peptide 40 and 42 (Ab40 and Ab42) in CSF, following single oral doses of GSI-953, an investigational drug, in healthy young subjects and patients with Alzheimer Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* For Healthy Young Subjects: Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and 12 lead ECGs.
* For AD patients: Patients must be generally healthy with the exception of Alzheimer Disease. (same as above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
We will assess the pharmacodynamics (PD) of biomarkers amyloid beta 40 and 42 in CSF, following single oral doses of GSI-953 in healthy young and Alzheimer's Patients. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Glendale, California, United States